CLINICAL TRIAL: NCT06374407
Title: Exploring the Interplay Between Diet, Obesity, Mental Health, and the Gut Microbiome. The MIND-GUT Digital Pilot Intervention Study.
Brief Title: The MIND-GUT Digital Pilot Intervention Study
Acronym: MINDGUT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Skövde (Other)
Collaborators: State University of New York - Downstate Medical Center (Other); Albert Einstein College of Medicine (Other); Göteborg University (Other); Uppsala University (Other); Kristianstad University (Other); University of Pavia (Other); The Food Scientist AB (Sweden) (Unknown)
Responsible Party: Principal Investigator, Gianluca Tognon, Senior lecturer in public health sciences, University of Skövde
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GT-001
Record Dates: First submitted 2024-04-04; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Obesity; Depressive Symptoms; Anxiety; Stress; Eating Habit; Dysbiosis
Keywords: mental health; obesity; mind gut diet; gut microbiome
MeSH Terms: conditions — Obesity; Depression; Anxiety Disorders; Feeding Behavior; Dysbiosis; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: We plan to randomly assign participants to either the intervention or control group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be blinded to their group assignment and will use a smartphone app for meal planning. However, those in the intervention group may have some awareness of their assignment due to specific food choices. Meanwhile, the control group will have access to a variety of foods and recipes, maintaining blinding between the groups regarding their assigned diets, addressing a common challenge in diet intervention studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): The control group comprises participants who do not receive the specific Mind diet intervention but undergo the same procedures as the intervention group, including weighing at the beginning and end of the study, completing identical questionnaires, and providing fecal samples at recruitment and follow-up. They will also use the same meal-planning app as the intervention group.
  Interventions: Behavioral: Dietary intervention based on the MIND diet
- Intervention group (Experimental): The intervention group consists of participants who receive the Mind diet intervention. Like the control group, they will be weighed at the start and end of the study, answer the same questionnaires, and provide fecal samples at recruitment and follow-up. Additionally, they will use the same meal-planning app as the control group, but their dietary pattern will be based on the Mind diet.
  Interventions: Behavioral: Dietary intervention based on the MIND diet

INTERVENTIONS:
Behavioral: Dietary intervention based on the MIND diet — A 12-week pilot randomized controlled trial (RCT) involving N=126 obese participants (1:1 gender ratio) to assess protocol feasibility, including recruitment, retention, compliance, physical examinations, and gut sample collection. Sample size, calculated by a statistician, expects a 5% body weight change at follow-up (std. dev. 10%). We chose a 12-week duration for this pilot study to allow sufficient time to observe significant changes in both body weight and mental health.

SUMMARY:
This 12-week pilot study aims to evaluate the feasibility and effectiveness of a dietary intervention targeting diet, obesity, mental health, and the gut microbiome in promoting weight loss and enhancing mental health among obese men and women aged 30-50. Participants, excluding those with specific medical conditions, will be randomly assigned to either an intervention or control group using a meal planning smartphone app. Clinical assessments will include anthropometry, mental health questionnaires, dietary recalls, and stool sample collections. The study's endpoints include program retention, adherence, changes in body weight, mental health, and gut microbiome diversity. Statistical analyses will evaluate intervention effects and the potential mediating roles of the gut microbiome. This pilot study has implications for health policies, public healthcare, digital health companies, and the biotech and pharmacology industries. Future plans involve a large-scale intervention study in multiple countries with ongoing collaborations.

DETAILED DESCRIPTION:
Objective of the Pilot Study and Study Design:

This 12-week randomized pilot intervention study aims to assess the feasibility and effectiveness of a dietary intervention targeting diet, obesity, mental health, and the gut microbiome in promoting weight loss and enhancing mental health among obese individuals aged 30-50.

Participant Recruitment and Randomization:

Participants aged 30-50, excluding those with specific medical conditions such as psychiatric medication use, food allergies affecting diets, eating disorders, diabetes, polycystic ovary syndrome, sensory deficits, recent antibiotic use, participation in other studies, language limitations, coeliac/inflammatory bowel disease, planned weight management within 3 months, and pregnant/lactating/post-menopausal women, will be recruited for the study. Randomization will be conducted to assign eligible participants to either an intervention or control group using a meal planning smartphone app.

Clinical Assessments:

Clinical assessments will include anthropometry, mental health questionnaires, dietary recalls, and stool sample collections.

Study Endpoints:

The study's endpoints include program retention, adherence, changes in body weight, mental health, and gut microbiome diversity.

Statistical Analyses:

Statistical analyses will evaluate the study feasibility, intervention effects on body weight and mental health changes, and the potential mediating roles of these effects by the gut microbiome.

Implications and Future Plans:

This pilot study has implications for health policies, public healthcare, digital health companies, and the biotech and pharmacology industries. Future plans involve a large-scale intervention study in multiple countries with ongoing collaborations.

ELIGIBILITY:
Inclusion Criteria:

* age 30- 50;
* BMI ≥ 30 kg/m2;
* stable physical activity;
* one person per household;
* commitment to full protocol.

Exclusion Criteria:

* use of psychiatric medications (e.g., serotonin reuptake inhibitors);
* use of weight loss medications (GLP-1 receptor agonists);
* food allergies affecting adherence to the MIND diet;
* diagnosis of eating disorders;
* diagnosis of diabetes;
* diagnosis of polycystic ovary syndrome;
* sensory deficits (e.g., COVID-19-induced loss of taste/smell);
* antibiotic use during the latest 3 months;
* participation in another study;
* language understanding limitations (i.e., not able to understand either Swedish or English); - coeliac/inflammatory bowel disease;
* planned weight management program within three months;
* pregnancy;
* lactation;
* menopause.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Program retention | 12 weeks
  Evaluation of participants' continued engagement in the program over time i.e., % of individuals completing the second and third 24h diet recall and % of participants returning to the second visit at the end of the intervention.
Adherence | 12 weeks
  Measurement of participants' compliance with the assigned diet and program through 24h recall interviews, assessed comparing reported intake frequencies of each food group with the recommended intake frequencies according to the principles of the MIND diet.
Acceptability | 12 weeks
  Assessment of participants' experience of the program through qualitative interviews, focusing in particular on: Perception of and experience with the intervention, intervention components (dietary plans, use of the app, etc.), factors influencing participants' engagement, perceived impact on behavior and well-being, interaction with the staff, suggestions for improvement.
Study effectiveness: change in eating attitudes at follow-up | 12 weeks
  Comparison of a score calculated after administration of the EAT-26 questionnaire at baseline vs. follow-up. The EAT-26 comprises three subscales, namely, Dieting, Bulimia and Food Preoccupation, and Oral Control. Higher scores correspond to a worse outcome.
Study effectiveness: change in stress levels at follow-up | 12 weeks
  Comparison of PSS-4 questionnaire at baseline vs. follow-up. The PSS total score is calculated by reverse-coding the positive items and summing the scores for all items. The total scores range from 0 to 56, from 0 to 40, and from 0 to 16 for the PSS-14, PSS-10, and PSS-4, respectively. A higher score indicates more perceived stress.
Study effectiveness: change in depression symptoms at follow-up | 12 weeks
  Comparison of PHQ-9 questionnaire at baseline vs. follow-up. The PHQ-9 is a tool to assist clinicians in identifying and diagnosing major depression. It has a maximum score of 27. Higher scores correspond to worst outcomes in terms of depression symtoms.
Study effectiveness: change in anxiety symtoms at follow-up | 12 weeks
  Comparison of GAD-7 questionnaire at baseline vs. follow-up. Each item is scored on a four-point Likert scale (0-3) with total scores ranging from 0 to 21 with higher scores reflecting worst outcomes in terms of anxiety severity.
Study effectiveness: change in body weight at follow-up | 12 weeks
  Comparison of body weight at baseline vs. follow-up
Study effectiveness: change in % total fat mass at follow-up | 12 weeks
  Comparison of body % total fat mass at baseline vs. follow-up
Study effectiveness: change in % visceral fat mass at follow-up | 12 weeks
  Comparison of body % visceral fat at baseline vs. follow-up
Study effectiveness: change in waist circumference at follow-up | 12 weeks
  Comparison of waist circumference at baseline vs. follow-up
Study effectiveness: change in hip circumference at follow-up | 12 weeks
  Comparison of hip circumference at baseline vs. follow-up
Study effectiveness: change in microbiome variety at follow-up | 12 weeks
  Comparison of number and types of species at baseline vs. follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Skövde, Skövde, Sweden